CLINICAL TRIAL: NCT02842541
Title: An Open Label, Multi-Center, Safety Study of Intravitreal EBI-031, an Interleukin-6 (IL-6) Inhibitor, Administered as Single and Repeat Injections in Subjects With Diabetic Macular Edema (DME)
Brief Title: Safety Study of Intravitreal EBI-031 Given as a Single or Repeat Injection to Subjects With Diabetic Macular Edema
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: New study planned.
Sponsor: Eleven Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EBI-031-1
Record Dates: First submitted 2016-07-19; First posted 2016-07-25 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Diabetic Macular Edema

ARMS (2):
- Single dose arm (Experimental): Subjects will receive a single intravitreal dose of EBI-031
  Interventions: Drug: EBI-031
- Repeat dose arm (Experimental): Subjects will receive an intravitreal dose of EBI-031 monthly for 3 months
  Interventions: Drug: EBI-031

INTERVENTIONS:
Drug: EBI-031

SUMMARY:
The purpose of the study is to evaluate the safety, tolerability, immunogenicity, and pharmacokinetics of up to 3 dose levels of EBI-031 given as an intravitreal injection in subjects with diabetic macular edema. There are two arms to the study, a single dose arm (1 dose) and a repeat dose arm (1 dose each month for 3 months). Eligible subjects will initially enroll in the single dose arm and 3 to 6 subjects will be dosed at each of the 3 dose levels. Safety will be assessed over the 28 days after the single dose prior to moving to the next higher dose level. Once all subjects in the single dose arm have been dosed with EBI-031 and the safety has been assessed eligible subjects will begin enrolling in the repeat dose arm. Subjects in the repeat dose arm will receive one dose each month for 3 months and will be assessed for safety. Escalation to the next higher dose will occur once it is determined safe to proceed to the next dose level. Six subjects will be dosed at each of the 3 dose levels.

ELIGIBILITY:
Inclusion Criteria:

* Give written voluntary informed consent and any authorizations required by local law
* Have a diagnosis of Type 1 or 2 diabetes mellitus
* Have decreased vision determined primarily to be the result of DME in the study eye
* Mean central foveal thickness on Spectral Domain Ocular Coherence Tomography (SD-OCT)> 325 in the study eye within 2 weeks of dosing
* Have best corrected Early Treatment of Diabetic Retinopathy Study (ETDRS) letter score of <73 (~20/40) and >19 (~20/400) in the study eye within 2 weeks of dosing.

Exclusion Criteria:

* Female that is pregnant and lactating
* Any prior history of anti-interleukin 6 (anti-IL-6) treatment, for example: tocilizumab, sirukumab, sarilumab, olokizumab
* Any concurrent biologics for immune disease such as anti-tumor necrosis factor (TNF): Enbrel (etanercept), Humira (adalimumab), Remicade (infliximab); an anti-interleukin 12 (anti-IL-12): Stelara (ustekinumab); or an anti-interleukin 1 (anti-IL-1): Kineret (anakinra), Ilaris (canakinumab), Arcalyst (rilonacept).
* Unstable, uncontrolled diabetes defined as hemoglobin A1C (HbA1C)≥10.5% within 3 months prior to dosing of EBI-031
* Received intravitreal anti-vascular endothelial growth factor (anti-VEGF) such as Eylea (aflibercept) within 8 weeks, Lucentis (ranibizumab) and Avastin (bevacizumab) within 4 months prior to EBI-031
* Significant renal disease, liver disease, or acute congestive heart failure
* History of myocardial infarction (MI), stroke, or transient ischemic attack (TIA)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-09; Primary Completion 2017-10 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Safety, tolerability, and immunogenicity as measured by adverse events and anti-drug antibody development of single and repeat doses of EBI-031 | Measure over the 84 days
  Number of Participants With Abnormal Laboratory Values, Adverse Events, and/or antibodies to EBI-031

CONTACTS AND LOCATIONS:
Overall Officials: Karen Tubridy, Study Director — Eleven Biotherapeutics